CLINICAL TRIAL: NCT02421640
Title: A Study of Adoptive Immunotherapy With Autologous Tumor Infiltrating Lymphocytes and Concurrent Chemoradiotherapy in Nasopharyngeal Carcinoma
Brief Title: Phase II Trial of TIL Following CCRT in Patients With Locoregionally Advanced NPC
Acronym: TIL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hai-Qiang Mai,MD,PhD, Deputy Director of the Department of Nasopharyngeal Carcinoma, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NPC and TIL
Record Dates: First submitted 2015-04-11; First posted 2015-04-20 (Estimated); Last update posted 2016-10-18 (Estimated); Status verified 2016-09

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cisplatin+TIL (Experimental): Cisplatin concurrent chemoradiotherapy(CCRT) combined with tumor-infiltrating lymphocyte (TIL)
  Interventions: Drug: Cisplatin+TIL
- Cisplatin (Active Comparator): Cisplatin concurrent chemoradiotherapy(CCRT) only
  Interventions: Drug: Cisplatin

INTERVENTIONS:
Drug: Cisplatin+TIL — cisplatin 100mg/m2(every three weeks),D1,D22,D43 of radiotherapy,then TIL infusing following concurrent chemoradiotherapy
  Other Names: DDP
  Arms: Cisplatin+TIL
Drug: Cisplatin — cisplatin 100mg/m2(every three weeks),D1,D22,D43 of radiotherapy only
  Other Names: DDP
  Arms: Cisplatin

SUMMARY:
This is a Phase II trial to study the effectiveness and security of cisplatin concurrent chemoradiotherapy plus TIL versus cisplatin concurrent chemoradiotherapy only with IMRT in treating patients with locoregionally advanced high risk nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
Nasopharyngeal carcinoma (NPC) is endemic in Southern China and Southeast Asia. For locoregionally advanced NPC,especially for the high risk NPC (EB virus DNA ≥ 4000 copies/ml) ,the incidence of treatment failure is still high. Although concurrent chemoradiotherapy (CCRT) can improve the treatment outcomes of these patients, approximately 25% of locoregionally advanced NPCs relapse. Adjuvant chemotherapy or inducing chemotherapy addition to CCRT did not significantly improve patient survival compared to CCRT alone. Hence, there is an urgent need for novel therapies to improve disease-free survival and reduce treatment-related toxicity in patients.

Accumulating evidence shows that tumor-infiltrating lymphocytes (TILs) selected for tumor recognition and greatly expanded in vitro are especially effective for treating cancer patients.The investigations phase I results showed that TILs following CCRT as a novel treatment strategy in locoregionally advanced NPC patients resulted in sustained anti-tumor activity and anti-EBV immune responses, associated with a good tolerance.

This is a Phase II trial to study the effectiveness and security of cisplatin CCRT plus TIL versus cisplatin CCRT only with IMRT in treating patients with locoregionally advanced high risk NPC.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly histologically confirmed non-keratinizing nasopharyngeal carcinoma, including WHO II or III
* Original clinical staged as T3-4N1-3 M0 or any T、N2-3M0（according to the 7th AJCC edition）
* No evidence of distant metastasis (M0)
* Plasm EB Virus DNA≥4000copies/ml
* Male and no pregnant female
* Satisfactory performance status: ECOG (Eastern Cooperative OncologyGroup) scale 0-1
* WBC ≥ 4×109 /L and PLT ≥4×109 /L and HGB ≥90 g/L
* With normal liver function test (ALT、AST ≤ 2.5×ULN, TBIL≤ 2.0×ULN)
* With normal renal function test (Creatinine ≤ 1.5×ULN)

Exclusion Criteria:

* Patients have evidence of relapse or distant metastasis
* Histologically confirmed keratinizing squamous cell carcinoma (WHO I)
* Receiving radiotherapy or chemotherapy previously
* The presence of uncontrolled life-threatening illness
* Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant.
* Active systemic infections, coagulation disorders or other major medical illnesses of the cardiovascular, respiratory or immune system, myocardial infarction, cardiac arrhythmias, obstructive or restrictive pulmonary disease.
* Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
* Concurrent opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities).
* Concurrent systemic steroid therapy
* HIV positive
* Suffered from other malignant tumors (except the cure of basal cell carcinoma or uterine cervical carcinoma in situ) previously

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2015-03; Primary Completion 2017-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Progress-free survival | 3 years
  Progress-free survival is calculated from the date of randomization to the date of the first progress at any site.

SECONDARY OUTCOMES:
Overall Survival (OS) | 3 years
  The OS was defined as the duration from the date of random assignment to the date of death from any cause or censored at the date of the last follow-up.
Locoregional Relapse-Free Survival (LRRF) | 3 years
  The LRRFS is evaluated and calculated from the date of random assignment until the day of first locoregional relapse or until the date of the last follow-up visit.
Distant Metastasis-Free Survival (DMFS) | 3 years
  The DMFS is evaluated and calculated from the date of random assignment until the day of first distant metastases or until the date of the last follow-up visit.
Complete Response (CR) | after the completion of the chemoradiotherapy treatment (up to 9 weeks)
  CR assessed by independent reviewers, according to the Modified Response Evaluation Criteria in Solid Tumors (RECIST) from the National Cancer Institute (NCI). Disease response evaluated after the completion of the chemoradiotherapy treatment. Complete response defined as the complete disappearance of the target and non-target lesion(s) identified at baseline after radiological evaluation by Magnetic Resonance Imaging (MRI) only.
Determine the toxic effects in these patients. | 4 weeks
  Patients will be monitored for clinical toxicity by standard NIH criteria. A time period of 4 weeks will constitute the time for clinical safety monitoring.
Determine the molecular expression of EBV DNA. | 12 weeks
  The molecular expression responses of the patients, including their plasma EBV DNA load, IFN levels and the expansion of EBV-antigen specific T cells.
Determine the quality of life (QoL) of these regimens in these patients. | 4 weeks
  Administration and Monitoring Patients will be evaluated in the clinic and eligibility and informed consent obtained. QoL was assessed using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire C30 (EORTCQLQ-C30) and EORTC QLQ Head and Neck.

CONTACTS AND LOCATIONS:
Overall Officials: Haiqiang Mai, MD,PhD, Principal Investigator — Cancer center
Locations (1):
- Haiqiang Mai, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided
decided by the results

REFERENCES:
- [Background] Chan AT, Leung SF, Ngan RK, Teo PM, Lau WH, Kwan WH, Hui EP, Yiu HY, Yeo W, Cheung FY, Yu KH, Chiu KW, Chan DT, Mok TS, Yau S, Yuen KT, Mo FK, Lai MM, Ma BB, Kam MK, Leung TW, Johnson PJ, Choi PH, Zee BC. Overall survival after concurrent cisplatin-radiotherapy compared with radiotherapy alone in locoregionally advanced nasopharyngeal carcinoma. J Natl Cancer Inst. 2005 Apr 6;97(7):536-9. doi: 10.1093/jnci/dji084. PMID 15812080
- [Background] Zhang L, Chen QY, Liu H, Tang LQ, Mai HQ. Emerging treatment options for nasopharyngeal carcinoma. Drug Des Devel Ther. 2013;7:37-52. doi: 10.2147/DDDT.S30753. Epub 2013 Feb 1. PMID 23403548
- [Background] Baujat B, Audry H, Bourhis J, Chan AT, Onat H, Chua DT, Kwong DL, Al-Sarraf M, Chi KH, Hareyama M, Leung SF, Thephamongkhol K, Pignon JP; MAC-NPC Collaborative Group. Chemotherapy in locally advanced nasopharyngeal carcinoma: an individual patient data meta-analysis of eight randomized trials and 1753 patients. Int J Radiat Oncol Biol Phys. 2006 Jan 1;64(1):47-56. doi: 10.1016/j.ijrobp.2005.06.037. PMID 16377415
- [Background] Chen L, Hu CS, Chen XZ, Hu GQ, Cheng ZB, Sun Y, Li WX, Chen YY, Xie FY, Liang SB, Chen Y, Xu TT, Li B, Long GX, Wang SY, Zheng BM, Guo Y, Sun Y, Mao YP, Tang LL, Chen YM, Liu MZ, Ma J. Concurrent chemoradiotherapy plus adjuvant chemotherapy versus concurrent chemoradiotherapy alone in patients with locoregionally advanced nasopharyngeal carcinoma: a phase 3 multicentre randomised controlled trial. Lancet Oncol. 2012 Feb;13(2):163-71. doi: 10.1016/S1470-2045(11)70320-5. Epub 2011 Dec 7. PMID 22154591
- [Background] Chen QY, Wen YF, Guo L, Liu H, Huang PY, Mo HY, Li NW, Xiang YQ, Luo DH, Qiu F, Sun R, Deng MQ, Chen MY, Hua YJ, Guo X, Cao KJ, Hong MH, Qian CN, Mai HQ. Concurrent chemoradiotherapy vs radiotherapy alone in stage II nasopharyngeal carcinoma: phase III randomized trial. J Natl Cancer Inst. 2011 Dec 7;103(23):1761-70. doi: 10.1093/jnci/djr432. Epub 2011 Nov 4. PMID 22056739
- [Background] Leung SF, Zee B, Ma BB, Hui EP, Mo F, Lai M, Chan KC, Chan LY, Kwan WH, Lo YM, Chan AT. Plasma Epstein-Barr viral deoxyribonucleic acid quantitation complements tumor-node-metastasis staging prognostication in nasopharyngeal carcinoma. J Clin Oncol. 2006 Dec 1;24(34):5414-8. doi: 10.1200/JCO.2006.07.7982. PMID 17135642
- [Background] Lin JC, Wang WY, Chen KY, Wei YH, Liang WM, Jan JS, Jiang RS. Quantification of plasma Epstein-Barr virus DNA in patients with advanced nasopharyngeal carcinoma. N Engl J Med. 2004 Jun 10;350(24):2461-70. doi: 10.1056/NEJMoa032260. PMID 15190138
- [Background] Louis CU, Straathof K, Bollard CM, Ennamuri S, Gerken C, Lopez TT, Huls MH, Sheehan A, Wu MF, Liu H, Gee A, Brenner MK, Rooney CM, Heslop HE, Gottschalk S. Adoptive transfer of EBV-specific T cells results in sustained clinical responses in patients with locoregional nasopharyngeal carcinoma. J Immunother. 2010 Nov-Dec;33(9):983-90. doi: 10.1097/CJI.0b013e3181f3cbf4. PMID 20948438
- [Background] Louis CU, Straathof K, Bollard CM, Gerken C, Huls MH, Gresik MV, Wu MF, Weiss HL, Gee AP, Brenner MK, Rooney CM, Heslop HE, Gottschalk S. Enhancing the in vivo expansion of adoptively transferred EBV-specific CTL with lymphodepleting CD45 monoclonal antibodies in NPC patients. Blood. 2009 Mar 12;113(11):2442-50. doi: 10.1182/blood-2008-05-157222. Epub 2008 Oct 29. PMID 18971421
- [Background] Smith C, Tsang J, Beagley L, Chua D, Lee V, Li V, Moss DJ, Coman W, Chan KH, Nicholls J, Kwong D, Khanna R. Effective treatment of metastatic forms of Epstein-Barr virus-associated nasopharyngeal carcinoma with a novel adenovirus-based adoptive immunotherapy. Cancer Res. 2012 Mar 1;72(5):1116-25. doi: 10.1158/0008-5472.CAN-11-3399. Epub 2012 Jan 26. PMID 22282657
- [Background] Dudley ME, Gross CA, Langhan MM, Garcia MR, Sherry RM, Yang JC, Phan GQ, Kammula US, Hughes MS, Citrin DE, Restifo NP, Wunderlich JR, Prieto PA, Hong JJ, Langan RC, Zlott DA, Morton KE, White DE, Laurencot CM, Rosenberg SA. CD8+ enriched "young" tumor infiltrating lymphocytes can mediate regression of metastatic melanoma. Clin Cancer Res. 2010 Dec 15;16(24):6122-31. doi: 10.1158/1078-0432.CCR-10-1297. Epub 2010 Jul 28. PMID 20668005
- [Derived] Liang YJ, Chen QY, Xu JX, Liu XF, Xia JC, Liu LT, Guo SS, Song B, Wang P, Li JB, Liu Q, Mo HY, Guo L, Sun R, Luo DH, He J, Liu YN, Nie CP, Tang LQ, Li J, Mai HQ. A phase II randomised controlled trial of adjuvant tumour-infiltrating lymphocytes for pretreatment Epstein-Barr virus DNA-selected high-risk nasopharyngeal carcinoma patients. Eur J Cancer. 2023 Sep;191:112965. doi: 10.1016/j.ejca.2023.112965. Epub 2023 Jul 5. PMID 37540921